CLINICAL TRIAL: NCT06243029
Title: Clinical Observational Study of Remote, Non-invasive, Multidomain Endpoints in Patients Recovering From Acute Decompensated Heart Failure
Brief Title: A Study to Assess Multidomain Endpoints of an ECG Patch
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1840M00072
Record Dates: First submitted 2023-10-02; First posted 2024-02-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute Decompensated Heart Failure;; Heart Failure;; ECG Patch
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected and analysed for standard clinical chemistry and haematology, NT-proBNP sample, high sensitivity Troponin sample.
  Urine will also be collected for uACR-urine albumin-creatinine ratio and urine sodium.
  Blood samples for biomarker research such as O-Link and Proteomics will also be collected. The analysis is not limited to these methods and can encompass other relevant approaches.
  DNA/RNA analysis will not be performed in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ECG Patch — Wearable ECG Patch designed to record and transmit physiological parameters to a mobile device or a data cloud. The device stores data locally in a memory cache designed for >96 hours of continuous data. It continuously records a one-lead ECG and has a three-axis accelerometer. On-board algorithms use those data to compute heart rate, heart rate variability, RR-interval, respiratory rate, and an activity level indicator. The company also provides optional arrhythmia detection and reporting services, the results of which may be delivered to healthcare professionals.

SUMMARY:
This study aims to evaluate the utility of a wearable heart monitoring patch that can be worn on the body to collect various measurements related to heart failure and develop a concept to potentially be used as a new measurement. It is crucial to test out new ways that make it easier to do research for new drugs and increase our chances of knowing how well they will work early on in the development process. Results from this study will be useful in planning future development programs for drugs aimed at treating patients with heart disease.

This study will be conducted in a single hospital, it is non-randomised (not chosen by chance), exploratory, study in the United Kingdom (University Hospitals of Leicester NHS Trust). It aims to involve up to 80 men and women recently admitted due to sudden, severe heart failure symptoms. Participants will be part of the study for about two months, with one hospital visit after discharge, as commonly done in heart failure centres.

* Visit 1 (Pre-Screening/Screening/Enrolment) will assess the participant's eligibility for participating in the study and for collecting data following hospitalisation for acute decompensated heart failure (ADHF). Participants will be trained and receive an ECG patch to wear from that moment onwards at home for a period of 4 to 7 days.
* Visit 2 (Follow-up visit) will be conducted approximately 6-8 weeks post Visit 1 and this will be the final study-related site visit. Participants will receive an ECG patch to wear at home for a second time for a period of 4 to 7 days.
* Visit 3 (Review of Medical Records). It is a review of the health status using medical records by the study team. The participant is not expected to attend the hospital for any appointments

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older
* Confirmed diagnosis of heart failure according to the latest ESC criteria
* Primary cause of hospitalisation due to decompensated heart failure
* Willing and able to complete all visits and assessments as per protocol
* Provision of signed and dated, written informed consent before any study-specific procedures.

Exclusion Criteria:

* Receiving renal replacement therapy
* Implanted cardiac (or other) device in-situ, cardiac pacemaker, defibrillator, or other implanted electronic devices or other ventricular assist device in situ
* Currently receiving chemotherapy
* Receiving end-of-life care
* Active severe infection: individuals with an active severe infection, as determined by the PI's clinical judgment, will not be eligible for study participation
* Hypersensitivity to patch adhesive/ materials in the patch
* Skin condition or damage that prevents wearing of the patch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be identified through review of hospital inpatient lists, conversations with healthcare providers and review of medical notes. Participants who meet the study eligibility criteria will be approached whilst still in the hospital but due to be discharged by the research team who will enquire whether they are interested in participating in the study.
  Up to 80 male and female participants over 18 years old will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Change in patch-measured variables between baseline and follow-up at 6-8 weeks (multiple variables) using the ECG patch. | 6-8 weeks

SECONDARY OUTCOMES:
Data completeness overall and per ECG patch variable, participant adherence, signal to noise ratio, day versus night assessment of quality using the ECG patch. | 6-8 weeks
Correlation between a change in ECG patch variables (multiple) and change in KCCQ at 6-8 weeks after discharge from hospital following admission for ADHF. | 6-8 weeks
Correlation between clinical parameters e.g. NT-pro BNP, KCCQ, BP, HR and the patch variables using data from Visit 1 (multiple comparisons). | 6-8 weeks
Correlation between change in NT-proBNP, BP, HR, body weight, peripheral oedema extent, NYHA class etc. and change in the patch variables (multiple comparisons). | 6-8 weeks
Correlation between change in one minute sit to stand test, frailty score, hand grip test and the change in patch variables (multiple comparisons). | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof Iain Squire, BSc MBChB MD, Principal Investigator — Glenfield Hospital, University Hospitals of Leicester NHS Trust; Dr Owais Dar, MD PhD, Principal Investigator — Royal Brompton & Harefield Hospitals,Guy's and St Thomas' Foundation Trust; Dr Joseph Cheriyan, MD PhD, Principal Investigator — Cambridge University Hospitals NHS Trust
Locations (3):
- United Kingdom (3):
  - Research Site, Cambridge
  - Research Site, Harefield
  - Research Site, Leicester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual participant-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home